CLINICAL TRIAL: NCT04001751
Title: Feasibility Study of the "SKYPE" Educational Project in Patients With Breast Cancer Treated With Hormonotherapy
Brief Title: Feasibility Study: Yoga Educational Project
Acronym: SKYPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PROICM 2018-02 SKY; 2018-A00208-47 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2019-06-07; First posted 2019-06-28 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer
Keywords: breast cancer; hormonotherapy; osteoarticular pain; yoga; therapeutic patient education
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Therapeutic educational postural yoga program (Experimental): Daily 15-min yoga sessions at home during 12 weeks. One 90-min yoga-therapeutic education session/week (during 6 weeks).
  Interventions: Behavioral: educational yoga program

INTERVENTIONS:
Behavioral: educational yoga program — Daily 15-min yoga sessions at home with the "Le guide du yoga" and the audio-guide, during 12 weeks.
  One 90-min yoga-therapeutic education session/week (during 6 weeks) given by a physical therapist trained to postural yoga.

SUMMARY:
As much as 45 to 60% of patients treated with hormonotherapy (HT) for breast cancer (BC) suffer from osteoarticular pain during treatment. Secondary effects have become a real issue because of their consequences on the patients' quality of life, but also on treatment efficacy and survival when they induce dose reduction or premature withdrawal of treatment.

Additional medicines (acupuncture, hypnosis, yoga) have become more and more popular these last years. 48 to 80% of patients with BC eventually choose them. A review comparing efficacy of various therapies to decrease osteoarticular pain concludes to a highest efficacy of anti-inflammatory treatments, paracetamol and yoga.

With this project, the investigators will assess the feasibility of a therapeutic yoga program with home practice for patients with breast cancer treated with hormonotherapy. The investigators will measure adhesion of the patients to perform yoga postures in an autonomous manner. Our study will also allow collection of data on the effect of such a program on quality of life, in view of setting-up an intervention study.

DETAILED DESCRIPTION:
Numerous initiatives have started in France, often associative. It is essential to evaluate in a rigorous manner, these therapies before making them part of the patient's care pathway.

Yoga has shown a real benefit in terms of pain reduction in patients with BC treated with HT. These osteoarticular pains are the secondary effect on which a physical therapeutic care can have a real benefit.

It thus appears innovative to complete this care with a therapeutic education program (TEP) in postural yoga which will enable patients to practice yoga postures at home by themselves. Yoga allows a large adaptation to pains expressed by each patient. It will favor the development of the feeling of control that they have in particular on their pain. participants will so improve the self-efficacy, the quality of life, and will reduce their fatigue and their pain. The patients involved have already lived major body transformations because of the disease and treatments. Yoga will help them put their lives together again, both physically and psychologically, and reclaim their body.

Studies have shown the short-term effects of yoga practice on anxiety, stress, pain and quality of life. Few rare studies have suggested that patients could add yoga practice at home to the supervised sessions, but these studies lacked therapeutic patient education. To date, to our knowledge, no data on the effect of the realization of yoga postures at home on increase of the patients' self-competency feeling are available in France. Also, the long-term effects of such programs need to be assessed.

The Montpellier Cancer Institute (ICM) has set-up 8 years ago yoga sessions for women with breast cancer, together with an association located in Montpellier.

With this study, the investigators will assess the feasibility of an educational yoga program given by a trained physical therapist in patients with beast cancer treated with hormonotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Non metastatic breast cancer
* Ongoing hormonotherapy, with no treatment modification in the 30 days before inclusion
* Osteoarticular pain ≥ 4 (resting or moving) on the VAS (Visual Analogue Scale)
* Previous treatment (surgery, chemotherapy or radiotherapy) ended at least 2 months before inclusion
* Informed patient and signed informed consent received
* Affiliation to a social security category

Exclusion Criteria:

* Chronic rheumatologic pain with specific care needed
* Yoga practice in the 3 months before inclusion
* Contra-indication or clinical state not allowing physical practice

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-08-31 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
proportion of patient compliance to the educational yoga program | 12 weeks
  Compliance will be posittive if 70% of daily sessions at home and 4 sessions out of the 6 therapeutic educational (TEP) sessions delivered in the center by a physical therapist are realised

SECONDARY OUTCOMES:
the patients' satisfaction towards the program | 12 weeks
  Satisfaction will be measured using the Likert scale (0 no satisfy to 10: strongly satisfy)
the induced self-competency feeling | 12 weeks
  self-competency feeling induced will be assessed using the GSES (General Self Efficacy-Schwarzer) questionnaire (10 questions - scale 1- not at all true to 4-totally true)
To assess quality of life by Quality of Life Questionnaire | 12 weeks
  Quality of life will be measured by EORTC QLQ-C30 (Quality of Life Questionnaire)
To assess quality of life by Quality of Life Questionnaire specify for Breast Cancer | 12 weeks
  Quality of life will be measured by EORTC QLQ-Br23 (Quality of Life Questionnaire specify for Breast Cancer)
To assess fatigue and stress | 12 weeks
  Fatigue and stress will be assessed using a Visual Analogous Scale (VAS) (0: no fatigue or no stress to 10 - maximum fatigue or stress)
Anxiety and depression prevalence | 12 weeks
  Anxiety and depression will be assessed by HADS (Hospital Anxiety and Depression Scale) questionnaire (7 questions about Anxiety and 7 questions about Depression)
Osteoarticular pain | 12 weeks
  osteoarticular pain will be assessed using a Visual Analogous scale (0: no pain to 10: maximum pain)
Forward-flexion flexibility | 12 weeks
  Forward-flexion flexibility is defined by the distance between the fingertips and the floor. It will be measured with a ruler.
Respiratory capacity | 12 weeks
  Respiratory capacity will be measured with a spirometer
Compliance to hormonotherapy treatment | 12 weeks
  Taking hormonotherapy treatments will be reported in a log-book by the patients.
Patient enrolment rate | at baseline
  The patient enrolment rate will be estimated (i.e. the proportion of patients giving their consent to participate in the study among eligible screened patients).
Reasons of non-participation to the study. | at baseline
  The reason of non-participation to the study (difficulty of coming, not concerning by the project, not interesting by the project, fatigue, other) will be reported by the patient to the doctor.

CONTACTS AND LOCATIONS:
Overall Officials: Kerstin FARAVEL, Study Chair — Institut du Cancer de Montpellier - Val d'Aurelle
Locations (1):
- Institut du Cancer de Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lintermans A, Van Asten K, Wildiers H, Laenen A, Paridaens R, Weltens C, Verhaeghe J, Vanderschueren D, Smeets A, Van Limbergen E, Leunen K, Christiaens MR, Neven P. A prospective assessment of musculoskeletal toxicity and loss of grip strength in breast cancer patients receiving adjuvant aromatase inhibitors and tamoxifen, and relation with BMI. Breast Cancer Res Treat. 2014 Jul;146(1):109-16. doi: 10.1007/s10549-014-2986-7. Epub 2014 May 11. PMID 24816806
- [Background] Peppone LJ, Janelsins MC, Kamen C, Mohile SG, Sprod LK, Gewandter JS, Kirshner JJ, Gaur R, Ruzich J, Esparaz BT, Mustian KM. The effect of YOCAS(c)(R) yoga for musculoskeletal symptoms among breast cancer survivors on hormonal therapy. Breast Cancer Res Treat. 2015 Apr;150(3):597-604. doi: 10.1007/s10549-015-3351-1. Epub 2015 Mar 27. PMID 25814054
- [Background] Crew KD, Greenlee H, Capodice J, Raptis G, Brafman L, Fuentes D, Sierra A, Hershman DL. Prevalence of joint symptoms in postmenopausal women taking aromatase inhibitors for early-stage breast cancer. J Clin Oncol. 2007 Sep 1;25(25):3877-83. doi: 10.1200/JCO.2007.10.7573. PMID 17761973
- [Background] Greenlee H, Balneaves LG, Carlson LE, Cohen M, Deng G, Hershman D, Mumber M, Perlmutter J, Seely D, Sen A, Zick SM, Tripathy D; Society for Integrative Oncology. Clinical practice guidelines on the use of integrative therapies as supportive care in patients treated for breast cancer. J Natl Cancer Inst Monogr. 2014 Nov;2014(50):346-58. doi: 10.1093/jncimonographs/lgu041. PMID 25749602
- [Background] Lombard JM, Zdenkowski N, Wells K, Beckmore C, Reaby L, Forbes JF, Chirgwin J. Aromatase inhibitor induced musculoskeletal syndrome: a significant problem with limited treatment options. Support Care Cancer. 2016 May;24(5):2139-2146. doi: 10.1007/s00520-015-3001-5. Epub 2015 Nov 10. PMID 26556210
- [Result] Faravel K, Huteau ME, Jarlier M, de Forges H, Meignant L, Senesse P, Norton J, Jacot W, Stoebner A. Importance of Patient Education for At-home Yoga Practice in Women With Hormonal Therapy-induced Pain During Adjuvant Breast Cancer Treatment: A Feasibility Study. Integr Cancer Ther. 2021 Jan-Dec;20:15347354211063791. doi: 10.1177/15347354211063791. PMID 34939444